CLINICAL TRIAL: NCT05731037
Title: Patellar Tendinopathy - The Role of Restitution Time in Exercise- Based Treatment: A Randomized Controlled Trial (the TEREX Trial)
Brief Title: Influence of Restitution Time in Treatment of Patellar Tendinopathy
Acronym: TEREX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Anne-Sofie Agergaard, Postdoc, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The TEREX trial
Record Dates: First submitted 2023-01-27; First posted 2023-02-16 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Patellar Tendinopathy; Jumper's Knee
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short restitution group (SR) (Active Comparator): Resistance training for knee extensors three training session per week.
  Interventions: Other: Resistance training for knee extensors
- Extended restitution group (ER) (Experimental): Resistance training for knee extensors on training session per week (greater restitution from loading).
  Interventions: Other: Resistance training for knee extensors

INTERVENTIONS:
Other: Resistance training for knee extensors — The exercise will be started at 60% of 1 repetition maximum (RM) and progressed to 75% of 1 RM during the first 3 weeks and maintained throughout the intervention period. The exercise will be performed slowly (6 s/ repetition).

SUMMARY:
The purpose of the present project is to investigate if the restitution time from loading in an exercise-based 12 weeks rehabilitation regime for patellar tendinopathy influences the clinical outcome, tendon structure and function.

The investigators hypothesize that greater restitution from loading (1 exercise day per week) will yield a greater positive clinical outcome, and tissue structure and function in patients with patellar tendinopathy compared to less restitution (3 exercise days per week), when impact activities are restricted in both groups.

DETAILED DESCRIPTION:
This study is designed as a prospective, randomized, controlled, open label, superiority trial with a two-group parallel design and primary endpoint after 12 weeks. The study has two phases; The first phase includes the main trial in which a 12-week intervention period will be undertaken to test the hypotheses in patients with chronic patellar tendinopathy (symptoms > 3 months).

At 12 weeks, a smaller group of patients (responding and not-responding to the 12-week intervention period) will be offered to participate in sub-study 1. In this explorative cross-sectional study, the feasibility of mapping brain structure, function and metabolism using Magnetic resonance imaging (MRI) with Blood Oxygenation Level Dependent (BOLD) imaging technique in chronic patellar tendinopathy patients will be assessed.

The second phase in the main study includes the follow-up from 12 week to the secondary endpoint at 52 weeks after baseline. During this period the participants will be monitored via questionnaires for treatment satisfaction and improvements at 4-week intervals. What treatment and the duration of treatment patients will receive in this phase is based on the concept of personalized medicine. We expect the majority of patient to continue in the group with loading-based intervention. A smaller group of the 52 patients from the main study is expected to be included in sub-study two.

Sub study two is designed as an observational cohort study. In this sub study, patients reporting no self-evaluated improvement after 12 weeks of loading-based treatment will be asked to be part of a group receiving corticosteroid injection treatment followed by continued exercise-based treatment and avoidance of impact loading. The cohort will further include patients that after week 20, 24, 28, 32, 36 and 40 respond that they have not achieved their Patient Acceptable Symptom State (PASS).

ELIGIBILITY:
Inclusion Criteria:

* Sports active men and women.
* Age (18-60) years old.
* BMI (18.5-30)
* Understand and read Danish
* Uni- or bilateral patellar tendinopathy
* Symptom onset >90 days ago

Exclusion Criteria:

* Patellar tendinopathy longer than 24 months
* Smoking
* Previous surgery in the knee on the ipsilateral side.
* Corticosteroid injection in the patellar tendon on the ipsilateral side within the last 6 months.
* Any confounding diagnosis to the knee joint
* Known arthritis
* Known diabetes
* Inability to follow rehabilitation or complete follow-ups
* Enrolled in a resistance based-rehabilitation program for the affected patellar tendon within the previous three month
* Have a work were it is not feasible to avoid pain provoking tasks

Extra criteria sub-study one

Inclusion criteria:

• Five patients from the main study, rating "improved" and "not improved" respectively, will be invited to participate in sub-study one.

Exclusion criteria:

* Claustrophobia
* Pregnancy
* Breastfeeding

Extra criteria sub-study two:

Inclusion criteria:

* Patients from the main study, that rate themselves 'not improved' in symptoms after 12 week.
* Patients who have not achieved Patient Acceptable Symptom State (PASS) after week 20, 24, 28, 32, 36 and 40, will be invited to participate in sub- study two.

Exclusion criteria:

* Pregnancy
* Breastfeeding
* Previously had an allergic reaction for steroid (Depomedrol).
* Previously had an allergic reaction for local anesthesia treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-02-10 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Patient perception VISA-P | Change from baseline at week 12
  Change in Victorian Institute of Sports Assessment - patella (VISA-P) total score. The VISA-P asses symptoms, function and the ability to participate in sport. It consists of 8 questions, with a maximum score of 100 indicating the person is asymptomatic and fully per-forming and lower scores indicating more symptoms and limitations of function and activity.

SECONDARY OUTCOMES:
Patient perception VISA-P secondary | Change from baseline at week 16 and 52
  Change in Victorian Institute of Sports Assessment - patella (VISA-P) total score. The VISA-P asses symptoms, function and the ability to participate in sport. It consists of 8 questions, with a maximum score of 100 indicating the person is asymptomatic and fully per-forming and lower scores indicating more symptoms and limitations of function and activity.
Patient perception VISA-P truncated | Change from baseline at week 12, 16 and 52
  Change in Victorian Institute of Sports Assessment - patella (VISA-P) truncated score. The truncated score only including questions 2-6, with a maximum score of 50. Lower scores indicating more symptoms and limitations of function and activity.
Self-reported pain (NRS) - Preferred sport | Change from baseline at week 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52.
  Change in pain rating on an 11 point numeric rating scale (NRS) during preferred sport, with 10 being the worst imaginable pain and 0 denoting no pain.
Self-reported pain (NRS) - Rest | Change from baseline at week 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52.
  Change in pain rating on an 11 point numeric rating scale (NRS) during rest, with 10 being the worst imaginable pain and 0 denoting no pain.
Self-reported pain (NRS) - Daily activities | Change from baseline at week 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52.
  Change in pain rating on an 11 point numeric rating scale (NRS) during daily activities, with 10 being the worst imaginable pain and 0 denoting no pain.
Self-reported improvement (GROC) | Change from baseline at week 12, 16 and 52.
  Self-reported improvement after treatment will be evaluated by the Global Rating of change (GROC) on a 7-point Likert scale ranging from 'much improved' to 'much worse'.
Sports participation | Week 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52.
  Number of sports participation hours per week (training and competition).
Sports types | Week 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52.
  Typer of sports performed.
Sports intensity | Week 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52.
  Intensity of sport performed registred in a self-reported questianaire and categorized as; light, moderate or vigorous.
Self-reported satisfaction (PASS) | Week 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
  Self-evaluated satisfaction with treatment result will be evaluated by Patient Acceptable Symptom State (PASS) on a 5-point Likert scale ranging from 'very satisfied' to 'very unsaticfied'
Treatment received | Week 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52.
  Registration of any additive treatment received from last follow-up measured with self-reported questionnaire.
Care-seeking behavior | Week 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52.
  Registration of any additive care-seeking behavior from last follow-up measured with self-reported questionnaire.
The single-leg decline squat (SLDS) will be used to assess pain during function | Change from baseline at week 12 and 52.
  Participants performed a decline squat on a 25°decline board and reported pain using an 11 point numeric rating scale (NRS) upon completion, with 10 being the worst imaginable pain and 0 denoting no pain.
Muscle strength | Change from baseline at week 12 and 52.
  Maximal muscle strength is obtained during standardized maximal voluntary contractions.
Ultrasonography - tendon thickness | Change from baseline at week 12 and 52.
  Grey scale ultrasonography will be used for evaluation of patellar tendon thickness.
Ultrasonography - tendon neovascularization | Change from baseline at week 12 and 52.
  Doppler ultrasonography will be used for evaluation of patellar tendon neovascularization.
Ultrasonography - tendon microvascularisation | Change from baseline at week 12 and 52.
  B-Flow ultrasonography will be used for evaluation of patellar tendon microvascularisation.
Counter movement Jump height | Change from baseline at week 12 and 52.
  Jump height during Counter movement Jump test will be used to assess patellar tendinopathy caused functional deficits.

OTHER OUTCOMES:
Magnetic resonance imaging (MRI) with Blood Oxygenation Level Dependent (BOLD) imaging technique - Brain structure mapping. | At 12 weeks
  It will be testet If it is feasible to map brain structure changes in patient with chronic patellar tendinopathy using MRI BOLD imaging technique. The outcome will only be used for participants included in sub-study one.
Magnetic resonance imaging (MRI) with Blood Oxygenation Level Dependent (BOLD) imaging technique - Brain function mapping. | At 12 weeks
  It will be testet If it is feasible to map brain function changes in patient with chronic patellar tendinopathy using MRI BOLD imaging technique. The outcome will only be used for participants included in sub-study one.
Magnetic resonance imaging (MRI) with Blood Oxygenation Level Dependent (BOLD) imaging technique - Brain metabolism mapping. | At 12 weeks
  It will be testet If it is feasible to map brain metabolism changes in patient with chronic patellar tendinopathy using MRI BOLD imaging technique. The outcome will only be used for participants included in sub-study one.
Correlation between patient self-reported satisfaction and brain structure changes. | At 12 weeks
  Patient self-reported satisfaction will be assessed by Patient Acceptable Symptom State (PASS) and brain structure by Magnetic resonance imaging (MRI) with Blood Oxygenation Level Dependent (BOLD) imaging technique. The outcome will only be used for participants included in sub-study one.
Correlation between patient self-reported satisfaction and brain function changes. | At 12 weeks
  Patient self-reported satisfaction will be assessed by Patient Acceptable Symptom State (PASS) and brain function by Magnetic resonance imaging (MRI) with Blood Oxygenation Level Dependent (BOLD) imaging technique. The outcome will only be used for participants included in sub-study one.
Correlation between patient self-reported satisfaction and brain metabolism changes. | At 12 weeks
  Patient self-reported satisfaction will be assessed by Patient Acceptable Symptom State (PASS) and brain metabolism by Magnetic resonance imaging (MRI) with Blood Oxygenation Level Dependent (BOLD) imaging technique. The outcome will only be used for participants included in sub-study one.
Number of corticosteroid injections received | week 12 to 52
  Number of injections received from week 12-52 for patients participating in sub-study two.
Tendon thickness after injection. | Change from 1. injection and at week 4 and 8 after the injection.
  Grey scale ultrasonography will be used for evaluation of patellar tendon thickness. Only for patients participating in sub-study two.
Tendon neovascularization after injection. | Change from 1. injection and at week 4 and 8 after the injection.
  Doppler ultrasonography will be used for evaluation of patellar tendon neovascularization. Only for patients participating in sub-study two.
Tendon microvascular blood flow after injection. | Change from 1. injection and at week 4 and 8 after the injection.
  B-Flow ultrasonography will be used for evaluation of patellar tendon microvascularisation. Only for patients participating in sub-study two.
Self-reported satisfaction after injection. | Change from 1. injection and at week 4 and 8 after the injection.
  Self-evaluated satisfaction with treatment result will be evaluated by Patient Acceptable Symptom State (PASS) on a 5-point Likert scale ranging from 'very satisfied' to 'very unsaticfied'Symptom State (PASS) scale.
Registration of pain rating on numeric rating scale (NRS) during injection. | Week 12 to 52
  Pain rating will be evaluated on an 11 point numeric rating scale (NRS) during injection, with 10 being the worst imaginable pain and 0 denoting no pain. Only for patients participating in sub-study two.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical & Occupational Therapy/ Institute of Sports Medicine, Bispebjerg Hospital, Copenhagen, NV, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT05731037/Prot_SAP_001.pdf